CLINICAL TRIAL: NCT04871841
Title: Study of Sputnik V COVID-19 Vaccination in Adults in Kazakhstan
Status: Completed | Type: Observational
Sponsor: Karaganda Medical University (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 128/36-21-23
Record Dates: First submitted 2021-05-01; First posted 2021-05-04 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Covid19; Vaccine Adverse Reaction
Keywords: Sputnik V; Gam-COVID-Vac; Vaccine safety; Vaccine reactogenicity; Vaccine immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — Gam-COVID-Vac vaccine; RAD5 protein, S cerevisiae

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sputnik V Vaccinees: Participants (healthy adults aged >=18) will receive rAd26-S prime at day 0 and rAd5-S boost at day 21.
  Interventions: Biological: Sputnik V

INTERVENTIONS:
Biological: Sputnik V — Participants will receive intramuscular (IM) injection of a single dose of rAd26-S and rAd5-S at day 0 and day 21, respectively.
  Other Names: rAd26-S; rAd5-S; Gam-COVID-Vac

SUMMARY:
This study will assess the safety, reactogenicity, and immunogenicity of Gam-COVID-Vac (Sputnik V) vaccine intended to provide acquired immunity against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) causing coronavirus disease 2019 (COVID-19). The vaccine contains two recombinant adenoviral vectors harbouring SARS-CoV-2 Spike gene. The vaccine will be administered intramuscularly on a 2-dose prime-boost schedule. Participants will be healthy adults aged greater than or equal to 18 years, voluntarily undergoing vaccination according to the guidelines of the Ministry of Healthcare of Kazakhstan.

DETAILED DESCRIPTION:
Sputnik V (Gam-COVID-Vac) is an adenoviral vector vaccine developed by The Gamaleya Research Institute of Epidemiology and Microbiology (Moscow, Russia), registered and approved by the Ministry of Healthcare of Kazakhstan. The vaccine incorporates two recombinant adenoviral (rAd) vectors, rAd5 and rAd26, harbouring SARS-CoV-2 Spike (S) gene.

Earlier Phase I/II clinical trials established that Sputnik V is safe and efficacious when given intramuscularly in two sequential doses, as a rAd26-S prime at day 0 followed by rAd5-S boost at day 21, at 1x10^11 particles per dose. The aim of the current study is to provide data on the safety, reactogenicity, and immunogenicity of Sputnik V in adults vaccinated in Kazakhstan using the established vaccination regimen. In addition, the effects of prior COVID-19 exposure on the vaccine safety, reactogenicity, and immunogenicity will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy (in the physician's clinical judgment and as confirmed by medical records, and physical examination at screening).
* Willing to give informed consent, and answer short questionnaires on past exposure to COVID-19 and post-vaccination reactogenicity.
* Willing to comply with the requirements of the protocol.

Exclusion Criteria:

* Participant shows signs of an acute illness (excluding minor illnesses such as diarrhea or mild upper respiratory tract infection).
* Participant has a positive laboratory-confirmed test result for SARS-CoV-2 infection at screening.
* Deemed by investigators to be unlikely to complete study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by invitation to volunteer at vaccination clinic sites.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Adverse Events (AEs) for 21 Days after First Vaccination | day 21
  Solicited AEs are pre-defined local (at the injection site) and systemic adverse events, for which participants are questioned. Solicited local AEs include injection site pain, redness, swelling, itching. Solicited systemic AEs include fatigue, headache, myalgia, chills, fever, joint pain, nausea, vomiting, diarrhea, abdominal pain, rash external to injection site.
Number of Participants with Solicited Adverse Events (AEs) for 42 Days after First Vaccination | day 42
  Solicited AEs are pre-defined local (at the injection site) and systemic adverse events for which participants are questioned. Solicited local AEs include injection site pain, redness, swelling, itching. Solicited systemic AEs include fatigue, headache, myalgia, chills, fever, joint pain, nausea, vomiting, diarrhea, abdominal pain, rash external to injection site.
Change in the Titres of Systemic SARS-CoV-2 Binding Antibodies | Up to 6 months
  The titres of SARS-CoV-2 binding antibodies measured in serum/plasma.

SECONDARY OUTCOMES:
Change in the Titres of Mucosal SARS-CoV-2 Binding Antibodies | Up to 6 months
  The titres of SARS-CoV-2 binding antibodies measured in mucosal (nasal) swabs.
Change in the Titres of Systemic SARS-CoV-2 Neutralizing Antibodies | Up to 6 months
  The titres of SARS-CoV-2 neutralizing antibodies measured in serum/plasma.
Change in the titres of Mucosal SARS-CoV-2 Neutralizing Antibodies | Up to 6 months
  The titres of SARS-CoV-2 neutralizing antibodies measured in mucosal (nasal) swabs.
Change in the concentration of systemic cytokines | Up to 6 months
  The levels of cytokines measured in blood plasma.
Difference in the study outcomes between participants with and without prior COVID-19 exposure. | Up to 6 months
  The reactogenicity and immunogenicity readouts will be compared between participants with and without prior COVID-19 exposure, as defined by the presence of SARS-CoV-2-reactive antibodies prior to vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Kadyrova, MD, PhD, Principal Investigator — Research Centre, Karaganda Medical University; Sergey Yegorov, PhD, Principal Investigator — McMaster University, Hamilton, Canada; Anar Turmukhambetova, MD/DMS, Study Chair — Karaganda Medical University
Locations (1):
- Karaganda Medical University, Karaganda, Kazakhstan

REFERENCES:
- [Background] Yegorov S, Goremykina M, Ivanova R, Good SV, Babenko D, Shevtsov A, MacDonald KS, Zhunussov Y; COVID-19 Genomics Research Groupon behalf of the Semey COVID-19 Epidemiology Research Group. Epidemiology, clinical characteristics, and virologic features of COVID-19 patients in Kazakhstan: A nation-wide retrospective cohort study. Lancet Reg Health Eur. 2021 May;4:100096. doi: 10.1016/j.lanepe.2021.100096. Epub 2021 Apr 16. PMID 33880458
- [Result] Kadyrova I, Yegorov S, Negmetzhanov B, Kolesnikova Y, Kolesnichenko S, Korshukov I, Akhmaltdinova L, Vazenmiller D, Stupina Y, Kabildina N, Ashimova A, Raimbekova A, Turmukhambetova A, Miller MS, Hortelano G, Babenko D. High SARS-CoV-2 seroprevalence in Karaganda, Kazakhstan before the launch of COVID-19 vaccination. PLoS One. 2022 Jul 27;17(7):e0272008. doi: 10.1371/journal.pone.0272008. eCollection 2022. PMID 35895743
- [Result] Yegorov S, Kadyrova I, Negmetzhanov B, Kolesnikova Y, Kolesnichenko S, Korshukov I, Baiken Y, Matkarimov B, Miller MS, Hortelano GH, Babenko D. Sputnik-V reactogenicity and immunogenicity in the blood and mucosa: a prospective cohort study. Sci Rep. 2022 Aug 1;12(1):13207. doi: 10.1038/s41598-022-17514-3. PMID 35915123